CLINICAL TRIAL: NCT06384924
Title: Pilot Study of Raman Spectroscopic Imaging for Skin Cancer
Brief Title: Raman Spectroscopy and Skin Cancer
Status: Recruiting | Type: Observational
Sponsor: Renee Farrell (Other)
Responsible Party: Sponsor-Investigator, Renee Farrell, Medical Physicist, Clinical Assistant Professor, Stony Brook University
Organization: Stony Brook University (Other)
Other Study IDs: SBU-RAMAN-SKINCANCER
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Skin Cancer; Basal Cell Carcinoma; Squamous Cell Carcinoma
MeSH Terms: conditions — Skin Neoplasms; Carcinoma, Basal Cell; Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Raman Spectroscopy
  Interventions: Device: Raman Spectroscopy handheld probe (EmVision, FL, USA); Device: Raman Spectroscopy laser source (Hubner Photonics Inc, CA, USA)

INTERVENTIONS:
Device: Raman Spectroscopy handheld probe (EmVision, FL, USA) — The probe is approximately the size of a pen or pencil. The handheld probe is connected to the laser source using a cable. The probe is placed in light contact with the skin. The features of the laser light after it bounces off the skin is collected. This measurement can allow us to see tissue characteristics. This is a single session that will take approximately 15 minutes.
Device: Raman Spectroscopy laser source (Hubner Photonics Inc, CA, USA) — This light source will create the laser light that will pass through the cable and through the handheld probe onto the skin.

SUMMARY:
The goal of this observational study is to find out if Raman Spectroscopy, a type of imaging, can be used to determine the size of skin cancer tumors. The main question it aims to answer is:

-Can Raman Spectroscopy help figure out how far a tumor spreads?

This study will take measurements using laser light from an experimental, handheld probe by lightly touching the skin.

DETAILED DESCRIPTION:
Radiation therapy is an alternative to surgery for localized tumors with excellent tumor control and cosmetic outcome. Raman Spectroscopy has potential to be a useful non-invasive, non-destructive, real-time, in-vivo tool for differentiation of cancerous vs. non-cancerous tissues. With this knowledge and future studies, this will ultimately guide skin brachytherapy more accurately and avoid unnecessary radiation to cosmetically and functionally important tissues including eyelid, nose, lips or skin folds.

The purpose of this study is to determine the feasibility of Raman Spectroscopy to identify microscopic infiltration extent of skin cancer beyond grossly visible tumor, using artificial intelligence methods of supervised and un-supervised machine learning algorithms, including pattern recognition, convolutional neural networks, k-means clustering and principal component analysis.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed skin cancer (either basal cell carcinoma or squamous cell carcinoma)
* Participants must plan to receive brachytherapy treatment for the skin cancer at the study site.
* Ability to provide consent to the study.

Exclusion Criteria:

* Patient belongs to a vulnerable population (Minors (under 18 years old), Adults unable to consent, prisoners).
* Lesions on the eyelid or in close proximity to the eye
* Pregnant women, or women of childbearing age who refuse pregnancy testing.
* Patient has pacemaker.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will include patients with confirmed skin cancer.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2027-02-13 (Estimated); Study Completion 2027-02-13 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Raman Spectroscopy to observe differences in Raman spectra between visible lesion, skin surrounding lesion and contralateral normal skin. | 1 year
  Collect the Raman spectroscopy data starting from the center of visible lesion moving outward and also contralateral normal skin. Observe the different spectra peak wavelengths and intensities, which correspond to different chemical composition of the tissue. The Raman Spectra has units of wavelength Raman shift (1/centimeter) on the horizontal axis and arbitrary units of intensity on the vertical axis.

SECONDARY OUTCOMES:
Compare the size of clinically defined margin and Raman-defined margin | 1 year
  After generating a sufficient model for predicting cancerous from non-cancerous tissue based on Raman spectra, compare the volume of the clinically defined margin (uniform 1-2 centimeter margin upon clinical discretion) to the Raman-defined margin. The Raman-defined margin will not be used for treatment. The volume is measured in cc (cubic centimeter).
Compare the dose delivered to surrounding critical structures when using clinically defined margin and Raman-defined margin | 1 year
  Radiation dose to the critical structures (e.g., eyes) from the plan using clinically defined margin (uniform 1-2 centimeter margin upon clinical discretion) will be collected. A second plan (not to be used for treatment) will be generated based on the Raman-defined margin. The dose to critical structures will be compared for both plans. The unit for dose will be centiGray (cGy).

CONTACTS AND LOCATIONS:
Overall Officials: Renee Farrell, Principal Investigator — Stony Brook Cancer Center
Locations (1):
- Stony Brook Hospital, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No